CLINICAL TRIAL: NCT00892931
Title: Phase 2 Study of Azixa (MPC-6827) for the Treatment of Patients With Recurrent Glioblastoma Multiforme
Brief Title: Phase 2 Study MPC-6827 for Recurrent Glioblastoma Multiforme
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Myrexis Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MPC-6827-019
Record Dates: First submitted 2009-05-03; First posted 2009-05-05 (Estimated); Last update posted 2011-10-14 (Estimated); Status verified 2011-10

CONDITIONS: Glioblastoma Multiforme
Keywords: Glioblastoma; Brain Neoplasms; Recurrence
MeSH Terms: conditions — Glioblastoma; Brain Neoplasms; Recurrence | interventions — verubulin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Azixa — 3.3 mg/m2 of Azixa administered by intravenous infusion over 2 hours once weekly for 3 consecutive weeks every 4 weeks (1 cycle = 4 weeks)
  Other Names: MPC-6827

SUMMARY:
The purpose of this study is to determine the safety and effectiveness of Azixa in patients with recurrent glioblastoma multiforme

ELIGIBILITY:
Inclusion Criteria:

* Have histologically proven malignant Glioblastoma Multiforme in first or second relapse
* Have failed prior Fractionated External Beam Cranial Irradiation or IMRT
* Be at least 18 years old and with a life expectancy ≥ 8 weeks or ≥ 4 weeks if failed prior Avastin therapy
* Have a Karnofsky performance status of ≥ 60
* Have adequate bone marrow function, liver function, and renal function before starting therapy

Exclusion Criteria:

* Have had more than two relapses
* Have had radiosurgery
* Have a cardiac ejection fraction < 50% by MUGA or ECHO
* Have Troponin-I elevated above the normal range
* Have an increasing steroid requirement
* Have MRI evidence at baseline of enlarging or clinically significant intratumor hemorrhage
* Have active stroke and/or transient ischemic attack not optimally managed
* Have active cardiovascular disease (e.g. sub-optimally managed angina, impending myocardial infarction, or uncontrolled hypertension)
* Be pregnant or breast feeding
* Have had prior hypersensitivity reaction to Cremophor EL
* Be HIV positive

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2009-04; Primary Completion 2011-07 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
To determine the progression-free survival (PFS) rate | Six 28-day cycles from start of therapy

SECONDARY OUTCOMES:
Overall survival | 36 months
Overall response rate | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Beelen, MD, Study Director — Myrexis Inc.; Lawrence Recht, MD, Principal Investigator — Stanford University
Locations (10):
- United States (10):
  - Barrow Neurological Institute, Phoenix, Arizona
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Stanford University, Stanford, California
  - Northwestern University, Chicago, Illinois
  - Tufts Medical Center, Boston, Massachusetts
  - Lahey Clinic, Burlington, Massachusetts
  - University of Massachusettes, Worcester, Massachusetts
  - Darthmouth -Hitchcock Medical Center, Lebanon, New Hampshire
  - Columbia University, New York, New York
  - SCCA/University of Washington, Seattle, Washington

REFERENCES:
- [Background] Sirisoma N, Pervin A, Zhang H, Jiang S, Willardsen JA, Anderson MB, Mather G, Pleiman CM, Kasibhatla S, Tseng B, Drewe J, Cai SX. Discovery of N-(4-methoxyphenyl)-N,2-dimethylquinazolin-4-amine, a potent apoptosis inducer and efficacious anticancer agent with high blood brain barrier penetration. J Med Chem. 2009 Apr 23;52(8):2341-51. doi: 10.1021/jm801315b. PMID 19296653
- [Background] Kasibhatla S, Baichwal V, Cai SX, Roth B, Skvortsova I, Skvortsov S, Lukas P, English NM, Sirisoma N, Drewe J, Pervin A, Tseng B, Carlson RO, Pleiman CM. MPC-6827: a small-molecule inhibitor of microtubule formation that is not a substrate for multidrug resistance pumps. Cancer Res. 2007 Jun 15;67(12):5865-71. doi: 10.1158/0008-5472.CAN-07-0127. PMID 17575155
- See also: Myriad Pharmaceuticals Inc. is a biopharmaceutical company focused on discovering, developing, and commercializing novel small molecule drugs that address severe medical conditions, including cancer and HIV infection. — http://www.myriadpharma.com